CLINICAL TRIAL: NCT00346008
Title: Genetic Epidemiologic Studies of Melanoma in Iceland
Brief Title: Studying Genes to Identify Melanoma in Patients in Iceland and Their Family Members
Status: Completed | Type: Observational
Sponsor: Iceland Genomics Corporation (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: NBCI-03-033-CM; NCI-06-C-N026; CDR0000551606 (Registry Identifier: PDQ (Physician Data Query)); NBCI-01-087-CM; 999906026; NCT00482534 (obsolete NCT alias)
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2008-12

CONDITIONS: Melanoma (Skin)
Keywords: melanoma; recurrent melanoma; stage I melanoma; stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Chromatography, High Pressure Liquid

INTERVENTIONS:
Genetic: mutation analysis
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying the genes expressed in samples of blood from patients with cancer and their family members may help doctors identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying genes to identify melanoma in patients in Iceland and their family members.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the feasibility of Iceland Genomics Corporation (UVS) to identify melanoma in multiple-case families, individuals with multiple tumors, and selected additional family members in Iceland.
* Assess the feasibility of mutation detection using sequencing and HPLC.
* Determine UVS' ability to create datasets with demographic, epidemiologic and molecular data.

OUTLINE: Participants and patients undergo blood collection and complete lifestyle questionnaires. All patients and population-based controls have DNA samples sequenced for MC1R. Demographic and epidemiologic data on all study participants is collected. Sequencing of the major melanoma susceptibility genes CFDKN2A, CDK4, and MC1R is also performed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients diagnosed with melanoma and selected family members are eligible to participate
* Must live in Iceland

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Feasibility to identify melanoma
Feasibility to detect mutation
Ability to create datasets

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Goldstein, PhD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Iceland Genomics Corporation, Reykjavik, Iceland